CLINICAL TRIAL: NCT06151626
Title: Linking From an Artificial-Intelligence Driven Assessment of Upper Extremity Motor Adaptation to a Novel Multisensory-Rhythmic Intervention in Geriatric Rehabilitation
Brief Title: A Novel Multisensory-Rhythmic Intervention in Geriatric Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-ER-111-482
Record Dates: First submitted 2023-11-20; First posted 2023-11-30 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Virtual Reality; Hand Mirror; Geriatric; Kinesiology, Applied
MeSH Terms: interventions — Feedback, Sensory; Respiration

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- virtual-reality based rhythmic skill training (Experimental): Participants wear VR headsets and Oculus Touch controllers and undergo rhythm skill training for a total of 35 minutes.
  Interventions: Other: virtual-reality based rhythmic skill training; Other: breathing and muscle relaxation exercises
- rhythmic skill training with visual feedback (Active Comparator): The rhythm skill training activities in this group are the same as the virtual reality-based system. Participants received 35 minutes of rhythm skill training presented through a computer interface
  Interventions: Other: rhythmic skill training with visual feedback; Other: breathing and muscle relaxation exercises
- strengthening group (Active Comparator): The patients receive an upper limb strengthening exercise program under the supervision of a therapist to ensure that the strengthening exercises are performed correctly. This includes: proprioceptive neuromuscular facilitation, resistance training, and tendon gliding exercises.
  Interventions: Other: strengthening group; Other: breathing and muscle relaxation exercises

INTERVENTIONS:
Other: virtual-reality based rhythmic skill training — Participants wear VR headsets and Oculus Touch controllers and undergo rhythm skill training for a total of 35 minutes.
  Arms: virtual-reality based rhythmic skill training
Other: rhythmic skill training with visual feedback — The rhythm skill training activities in this group are the same as the virtual reality-based system. Participants received 35 minutes of rhythm skill training presented through a computer interface
  Arms: rhythmic skill training with visual feedback
Other: strengthening group — Participants receive an upper limb strengthening exercise program under the supervision of a therapist to ensure that the strengthening exercises are performed correctly. This includes: proprioceptive neuromuscular facilitation, resistance training, and tendon gliding exercises.
  Arms: strengthening group
Other: breathing and muscle relaxation exercises — 5 minutes of breathing and muscle relaxation exercises

SUMMARY:
Human performance takes shape from the dynamic interaction between person, environment, and task. Goal-directed action is a complex task, which requires the elderly to adapt their motor response according to the environment constraints and task requirements to accomplish the task goal. Among age-related problems, motor control deficits are often the main problems which restricts the frail elderly from maintaining independence for activities of daily living. Therefore, to preserve the quality of life, motor function of the elderly must be taken into consideration, including early detection of motor control problems and development of appropriate intervention strategy for persons with either healthy or pathological brain aging. Rhythmic skill training which is a new mode of dual tasks using rhythmic cueing as an external agent for facilitating an automatized motor task. During training, rhythmic skill training can provide multi-component of sensory stimulation, strengthen motor planning and optimize motor execution, therefore, it will improve the motor performance for the elderly or patients with mild cognitive impairment. In addition, the neuroplastic changes related to sensory processing, selective attention, or working memory demands through music rhythm training can facilitate the cognitive function for the elderly which is a current trend of geriatric rehabilitation. Moreover, the advantage of virtual reality is that it provides important information related to knowledge of result, which can induce better motor and cognitive training effects. Therefore, this research project will focus on assessing and intervening motor adaptation of upper extremity for the healthy elderly and patients with mild cognitive impairment. The first purpose of the project will analyze the difference in efficiency of responsive and predictive grasping motor adaptation among the healthy young adults, healthy elderly and patients with mild cognitive impairment through a test of perturbation-based of pinch-holding-up-activity, and use artificial intelligence for more accurate classification for the grasp pattern of healthy young adults, elderly and patients with mild cognitive impairment. The second one is to verify the effects of virtual-reality based rhythmic skill training system on the motor adaptation capability of upper limb and cognition for the elderly and patients with mild cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Montreal Cognitive Assessment (MoCA) score of 23 or higher,
2. Clinical Dementia Rating (CDR) of 0 (for normal subjects) or 1 (for mild cognitive impairment subjects),
3. Healthy young participants aged between 20-39 years, healthy older adults and mild cognitive impairment participants aged between 65-85 years,
4. No skeletal, muscular, or neurological problems in the upper limbs in the past year, and
5. Sufficient visual acuity to complete the tasks.

Exclusion Criteria:

* Any subjects with significant mental illness, central nervous system disorders, or medical history

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in responsive grip behavior | baseline, 8 weeks and 16 weeks
  To evaluate change in amplitude of pinch force development or adaptation to perturbation through a test of perturbation-based of pinch-holding-up-activity

SECONDARY OUTCOMES:
Change in the results of Semmes-Weinstein monofilament test | baseline, 8 weeks and 16 weeks
  To evaluate change in touch-deep pressure threshold of hands using a set of 20 nylon monofilaments with Semmes-Weinstein monofilament test
Change in the result of Purdue pegboard test | baseline, 8 weeks and 16 weeks
  To evaluate change in hand dexterity of dominant hand, non-dominant and both hands with a timed-test
Change in the result of Minnesota manual dexterity test | baseline, 8 weeks and 16 weeks
  To evaluate change in gross motor coordination of upper limb of dominant hand and both hands with a timed placing and turning test
Change in the result of Weber Two-Point Discrimination Test | baseline, 8 weeks and 16 weeks
  To evaluate the change in sensibility of the hands
The change in the results of Mini-Mental Status Examination (MMSE) | baseline, 8 weeks and 16 weeks
  To evaluate the changes in cognitive function in an individual over time with The MMSE test
The change in the results of Digit Span (DS) subtest from the Wechsler Adult Intelligence Scale-4th | baseline, 8 weeks and 16 weeks
  To evaluate the change in working memory, mental manipulation, cognitive flexibility and attention in an individual over time with Digit Span (DS) subtest
The change in the results of Knox Cube Test-Revised (KCT-R) | baseline, 8 weeks and 16 weeks
  To evaluate the change in short-term memory and attention span in an individual over time with a performance test
The change in the results of Conners continuous performance test-3 | baseline, 8 weeks and 16 weeks
  To evaluate attention related problems in an individual over time with a performance test

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No